CLINICAL TRIAL: NCT00600327
Title: Carotid Artery Revascularization Using the Boston Scientific EPI Filter Wire EZ™ and the EndoTex™ NexStent™
Acronym: CABERNET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Cheryl Fontana, Boston Scientific
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2209
Record Dates: First submitted 2008-01-14; First posted 2008-01-24 (Estimated); Last update posted 2008-01-24 (Estimated); Status verified 2008-01

CONDITIONS: Transient Ischemic Attack; Thromboembolic Stroke; Stroke Prevention
Keywords: Stroke; thrombosis; thromboembolic; Transient Ischemic Attack; TIA
MeSH Terms: conditions — Ischemic Attack, Transient; Stroke; Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Device: EndoTex™ NexStent™; Device: Filter Wire EZ™

INTERVENTIONS:
Device: EndoTex™ NexStent™ — EndoTex™ NexStent™ is a flexible, fine mesh Nitinol stent used to treat patients that are at high risk of adverse events from carotid endarterectomy and require carotid revascularization of a target vessel that has a reference diameter between 4mm and 9mm and stenosis that is less than 30mm in length.
Device: Filter Wire EZ™ — EPI Fliter Wire EZ™ Embolic Protection System is indicated for use as a guide wire and embolic protection system to contain and remove embolic material (thrombus/debris) while performing angioplasty and stenting procedures in coronary saphenous vein bypass grafts and carotid arteries.

SUMMARY:
The primary objective of this study is to demonstrate the safety of the NexStent for treatment of carotid artery lesions undergoing stenting with adjunctive use of the FilterWire distal embolic protection device. The rates will be compared to an Objective Performance Criterion (OPC) derived from historic data from high-risk patients undergoing surgical intervention with Carotid endarterectomy. Patients included in this study are those at higher risk for complications associated with CEA.

ELIGIBILITY:
Inclusion Criteria:

* patient is greater than or equal to 18 years of age.
* Anticipated patient life expectancy is of at least one year from the date of the index procedure.
* Lesion is located in the common carotid artery (CCA) and/or the internal carotid artery (ICA) or the carotid bifurcation.
* Target vessel is the only vessel being treated at this intervention and the lesion is less than or equal to 30 mm and can be treated with a single stent.
* Vessel to be treated is between 4.0 mm and 9.0 mm in diameter.
* Patient can be either symptomatic or asymptomatic; Symptomatic: Stenosis must be greater than or equal to 50% as determined by angiogram and the patient has a history of stroke, TIA and/or amaurosis fugax in the hemisphere supplied by the target vessel within 180 days of the procedure.
* Patient can be either symptomatic or asymptomatic; Asymptomatic: Stenosis must be greater than or equal to 60% as determined by angiogram without any neurological symptoms.
* Distal vessel "landing zone" for placement of the FilterWire must be between 3.5 mm and 5.5 mm in diameter with visual angiographic recommendations as described in the IFU.
* Female patients with no childbearing potential or a documented negative pregnancy test (urine or blood) within 10 days of the index procedure.
* Patient (or their legal guardian) understands the nature of the procedure and has provided a signed informed consent using a form that has been reviewed and approved by the Investigational Review Board/Ethics Committee of the respective clinical site prior to the procedure. This will be obtained prior to participation in the study.
* Patient is willing to comply with the protocol requirements and return to the treatment center for all required clinical evaluations
* Patient must fulfill at least one of the following Class I: Unstable angina, LVEF less than 30%, CHF class III or class IV, dialysis dependent renal failure, severe COPD, requirement for staged CABG or valve replacement post carotid index procedure,Previous carotid endarterectomy with significant restenosis, total occlusion of the contralateral carotid artery, Previous radiation treatment to the neck or radical neck dissection, Target lesion is at or above the second vertebral body C2 or below the clavicle, Inability to extend the head due to cervical arthritis or other cervical disorders, Tracheostomy or tracheal stoma,Presence of laryngeal nerve palsy, Bilateral carotid artery stenosis as determined by angiography.
* If a patient does not meet Class I criteria, a patient must meet two of the follwing class II criteria: Patient is greater than or equal to 75 years of age, Myocardial infarction within previous 6 weeks, Requires staged peripheral vascular surgery (i.e. abdominal aortic aneurysm repair) or other major surgery post carotid index procedure, Two or more proximal or major diseased coronary arteries with greater than or equal to 70% stenosis that have not or cannot be revascularized.

Exclusion Criteria:

* Previously placed stent in target vessel.
* Total occlusion of target vessel (ICA or CCA).
* Angiographically visible thrombus.
* Carotid string sign (a tiny, long segment of contrast in the true lumen of the artery, aneurysmal pouch formation, and the distal location of the arteriopathy) with poor visualization of the distal vessel.
* Vertebrobasilar insufficiency symptoms only, without clearly identifiable symptoms referable to the targeted carotid artery.
* Vessel anatomy precluding use of stent system or distal protection system.
* Presence of carotid artery dissection.
* Requirement for staged CABG, valve replacement or abdominal aortic aneurysm procedure 30 days before or after the index procedure.
* Evidence of a major disabling stroke within the previous 30 days.
* Patient has an evolving stroke or has experienced a major stroke (NIHSS score greater than or equal to 15) within 3 months.
* History of intracranial hemorrhage within the past 12 months.
* Any condition that precludes proper angiographic assessment or makes percutaneous arterial access unsafe, e.g. morbid obesity, history of chronic hypertension that is not controlled by medical therapy.
* Contraindication to heparin, aspirin, clopidogrel (Plavix®), X-ray contrast or ticlopidine (Ticlid®)in cases of intolerance to clopidogrel.
* History of liver failure with elevated prothrombin time.
* History or current indication of bleeding diathesis or coagulopathy.
* Hgb <8 gm/dl (unless on dialysis), platelet count < 50,000, WBC >15,000, INR > l.5 (irreversible) or heparin-associated thrombocytopenia.
* Known cardiac sources of emboli not under treatment with anticoagulant therapy.
* Atherosclerotic disease involving adjoining vessels precluding safe placement of the guiding catheter or sheath.
* Planned treatment of non-target lesion within 30 days.
* Other abnormal angiographic findings that indicate the patient is at risk of a stroke due to a problem other that the target lesion, such as: ipsilateral arterial stenosis greater in severity than the target lesion, cerebral aneurysm, or arteriovenous malformation (AVM) of the cerebral vasculature.
* Dementia or confusion.
* The patient is enrolled in another study protocol.
* Patient may not participate in another investigational trial up to 12 months post-index procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Actual)
Dates: Start 2001-12; Primary Completion 2005-03 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Major clinical events at one-year defined as any death, stroke or myocardial infarction | 1 year
30-day event rate defined as any death, stroke or myocardial infarction less than or equal to 30-days post-procedure; plus the 31-day to 12-month event rate defined as any ipsilateral stroke including any death as a result of an ipsilateral stroke. | 1 year

SECONDARY OUTCOMES:
NexStent™ technical success | post surgery
FilterWire EZ™ technical success | post surgery
Overall system technical success | post surgery
Angiographic success | post procedure
Procedure Success | 24 hours post procedure
Restenosis | 1 year
Target vessel revascularization | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Fontana, BSN, Study Director — Boston Scientific Corporation; L. Nelson Hopkins, MD, Principal Investigator — Millard Filmore/Gates Hospital; Subbarao Myla, MD, Principal Investigator — Hoag Hospital
Locations (19):
- United States (15):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - El Camino Hospital, Mountain View, California
  - Hoag Hospital, Newport Beach, California
  - Oschner Clinic Foundation, New Orleans, Louisiana
  - Union Memorial Hospital, Baltimore, Maryland
  - Albany Medical College, Albany, New York
  - Millard Fillmore Gates Hospital, Buffalo, New York
  - Columbia - Weill Cornell Division of Vascular Surgery, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Carolina Medical Center, Charlotte, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Harrisburg Hospital, Harrisburg, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh (UPMC-Shadyside), Pittsburgh, Pennsylvania
  - Swedish Medical Center, Seattle, Washington
- Favaloro Institute, Buenos Aires, Argentina
- Germany (3):
  - Cardiovascular Center Bethanien, Germany, Frankfurt
  - Leipzig Heart Center, Leipzig
  - Sieburg Heart Center, Germany, Siegburg

REFERENCES:
- [Derived] Hopkins LN, Myla SV, Grube E, Eles G, Dave R, Jaff MR, Allocco DJ. Carotid artery revascularisation in high-surgical-risk patients with the NexStent and the FilterWire EX/EZ: 3-year results from the CABERNET trial. EuroIntervention. 2010 Apr;5(8):917-24. PMID 20542776